CLINICAL TRIAL: NCT03341442
Title: Are Posterior Hip Precautions Necessary? A Randomized, Controlled Study of Posterior Hip Precautions After Total Hip Arthroplasty
Brief Title: A Study of Posterior Hip Precautions After Total Hip Arthroplasty
Acronym: HIPPRECAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: University of Kentucky (Other); Andrews Institute Orthopaedics & Sports Medicine (Unknown)
Responsible Party: Principal Investigator, Matthew Dietz, MD, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1512934414
Record Dates: First submitted 2017-10-25; First posted 2017-11-14 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No hip precautions (Experimental): No hip precautions practiced after THA surgery
  Interventions: Procedure: No hip precautions
- Hip precautions (No Intervention): Hip precautions practiced per standard of care after THA surgery

INTERVENTIONS:
Procedure: No hip precautions — No hip precautions practiced after THA surgery
  Arms: No hip precautions

SUMMARY:
The purpose of this study is to perform a randomized controlled study to compare patients undergoing THA via a posterolateral approach to receive either standard of care post-surgery hip restrictions or to receive no restrictions. The investigators goal is to first complete a pilot study in which the investigators assess the short term dislocation rates 3-6 months and then continue to recruit into this study and follow these patients for a year to determine the 1 year risk for dislocation. The investigators also will compare the HOOS Jr. and VAS scores and time until free from walking aid. The research question is: Will the elimination of post operative posterior hip precautions increase the dislocation rate? The hypothesis is that the elimination of post operative hip precautions will not increase the dislocation rate.

DETAILED DESCRIPTION:
1. Participants at the following institutions (West Virginia University; The Andrews Institute; and University of Kentucky Healthcare Sports Medicine will be given an educational session regarding hip replacement and procedures to follow after total hip replacement at their History and Physical visit prior to elective total hip replacement surgery via a posterior approach. 2. Participants will be told of the study after their educational session. All their questions will be answered and they will be given the opportunity to consent for participation. 3. After consent, the participant will be randomized to a control group receiving Standard of Care (education) hip precautions or to a 'no hip precautions' group. The control group will be instructed to practice postoperative hip precautions they learned at their educational session; (standard of care) (no flexion > 90 degrees, no internal rotation, no adduction) for 6 weeks. The intervention group will be aware of the precautions but will be told not to practice them post-operatively. 4. The participants will be monitored per the surgeons' normal routine post-operatively, which includes notification to the surgeon if the subject returns to the hospital with any hip problems. 5. After the first three participants who were randomized to 'no precautions' have returned for their post-op visit at all sites, the DSMB will have a teleconference to discuss any adverse events including dislocations. If any of the first 3 participants dislocated the study will be stopped. 6. At six weeks the following will be recorded: time to elimination of walking aids, dislocation episodes requiring closed reduction, and need for revision surgery. If any of the first 3 intervention participants dislocated during the 6 week period, the study will be stopped. 7. The participants will be asked to complete the HOOS Jr. and VAS follow-up questions at 2-week, 6-week, 3 month, 6 month and one year post-operatively per standard of care follow-up. Participants will be asked to list any hip precautions practiced at these time frames. 8. If the participants fail to come for the standard of care follow up appointments, the research assistant will call the participants and ask the HOOS Jr. and VAS questionnaires over the phone and to list any hip precautions they practiced.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective, primary, osteoarthritic total hip arthroplasty via a posterolateral approach

Exclusion Criteria:

* < 18 years of age, cognitive disorders, neuromuscular spasticity disorders, femoral neck fractures, connective tissue disorders (ie Ehlers Danlos), alcohol abuse, dual mobility implant, constrained implants, pregnant or planning to become pregnant at time of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Dislocation Rate | up to 1 year post op
  Occurrence of dislocations will be compared between groups.

SECONDARY OUTCOMES:
HOOS, JR (hip disability and osteoarthritis outcome score for joint replacement) | up to 1 year post op
  Change in baseline score over time will be compared between groups. This is a six question form asked at Pre-op, 2 week, 6 week, 3-6 month, and 1 year post op
Visual Analog Scale (VAS) | up to 1 year post op
  Change in baseline Visual Analog Scale (VAS) over time will be compared between groups. This scale is from 0-100, where 100 is the best, evaluating the patients Health State and will be given at Pre-op, 2 week, 6 week, 3-6 month, and 1 year post op
Time free from walking aid | up to 1 year post op
  Time taken to be free from walking aids will be used to identify differences between groups. This will be evaluated by the provider at 6 weeks, 3/6 months, and 1 year post op
Hip Precautions Practiced | up to 6 week post-op
  Hip precautions practiced per patient postoperatively will be compared between groups to identify change in dislocation rates. Patients will be asked at 2 & 6 week post op what if any precautions they practiced.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Dietz, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine Department of Orthopaedics, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be available. Group data will be published.

REFERENCES:
- [Background] Austrailian Orthopaedic Association National Joint Replacement Registry., Annual Report. 2012
- [Background] Hummel MT, Malkani AL, Yakkanti MR, Baker DL. Decreased dislocation after revision total hip arthroplasty using larger femoral head size and posterior capsular repair. J Arthroplasty. 2009 Sep;24(6 Suppl):73-6. doi: 10.1016/j.arth.2009.04.026. Epub 2009 Jul 4. PMID 19577890
- [Background] Soong M, Rubash HE, Macaulay W. Dislocation after total hip arthroplasty. J Am Acad Orthop Surg. 2004 Sep-Oct;12(5):314-21. doi: 10.5435/00124635-200409000-00006. PMID 15469226
- [Background] Suh KT, Park BG, Choi YJ. A posterior approach to primary total hip arthroplasty with soft tissue repair. Clin Orthop Relat Res. 2004 Jan;(418):162-7. doi: 10.1097/00003086-200401000-00026. PMID 15043109
- [Background] Ali Khan MA, Brakenbury PH, Reynolds IS. Dislocation following total hip replacement. J Bone Joint Surg Br. 1981;63-B(2):214-8. doi: 10.1302/0301-620X.63B2.7217144.
- [Background] Khatod M, Barber T, Paxton E, Namba R, Fithian D. An analysis of the risk of hip dislocation with a contemporary total joint registry. Clin Orthop Relat Res. 2006 Jun;447:19-23. doi: 10.1097/01.blo.0000218752.22613.78. PMID 16741469
- [Background] Pellicci PM, Bostrom M, Poss R. Posterior approach to total hip replacement using enhanced posterior soft tissue repair. Clin Orthop Relat Res. 1998 Oct;(355):224-8. doi: 10.1097/00003086-199810000-00023. PMID 9917607
- [Background] Phillips CB, Barrett JA, Losina E, Mahomed NN, Lingard EA, Guadagnoli E, Baron JA, Harris WH, Poss R, Katz JN. Incidence rates of dislocation, pulmonary embolism, and deep infection during the first six months after elective total hip replacement. J Bone Joint Surg Am. 2003 Jan;85(1):20-6. doi: 10.2106/00004623-200301000-00004. PMID 12533567
- [Background] Schmidt-Braekling T, Waldstein W, Akalin E, Benavente P, Frykberg B, Boettner F. Minimal invasive posterior total hip arthroplasty: are 6 weeks of hip precautions really necessary? Arch Orthop Trauma Surg. 2015 Feb;135(2):271-274. doi: 10.1007/s00402-014-2146-x. Epub 2015 Jan 4. PMID 25556661
- [Background] Barnsley L, Barnsley L, Page R. Are Hip Precautions Necessary Post Total Hip Arthroplasty? A Systematic Review. Geriatr Orthop Surg Rehabil. 2015 Sep;6(3):230-5. doi: 10.1177/2151458515584640. PMID 26328242
- [Background] Restrepo C, Mortazavi SM, Brothers J, Parvizi J, Rothman RH. Hip dislocation: are hip precautions necessary in anterior approaches? Clin Orthop Relat Res. 2011 Feb;469(2):417-22. doi: 10.1007/s11999-010-1668-y. PMID 21076896
- [Background] Barrett WP, Turner SE, Leopold JP. Prospective randomized study of direct anterior vs postero-lateral approach for total hip arthroplasty. J Arthroplasty. 2013 Oct;28(9):1634-8. doi: 10.1016/j.arth.2013.01.034. Epub 2013 Mar 19. PMID 23523485
- [Background] Graves SC, Dropkin BM, Keeney BJ, Lurie JD, Tomek IM. Does Surgical Approach Affect Patient-reported Function After Primary THA? Clin Orthop Relat Res. 2016 Apr;474(4):971-81. doi: 10.1007/s11999-015-4639-5. Epub 2015 Nov 30. PMID 26620966